CLINICAL TRIAL: NCT02486952
Title: Open, Non-Interventional, Multicenter Trial of MabThera in Combination With CHOP (or CHOP-like) Chemotherapy in Patients With Aggressive B-Cell Lymphoma
Brief Title: MabThera (Rituximab) in Combination With CHOP (or CHOP-like) Chemotherapy in Patients With Aggressive B-Cell Lymphoma
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Collaborators: Serbian Lymphoma Group (Unknown)
Responsible Party: Sponsor
Other Study IDs: ML20390
Record Dates: First submitted 2015-06-29; First posted 2015-07-01 (Estimated); Results first posted 2016-02-22 (Estimated); Last update posted 2016-02-22 (Estimated); Status verified 2016-01

CONDITIONS: Lymphoma, Lymphoma, Large B-Cell, Diffuse, Non-Hodgkin's Lymphoma, Lymphoma, Non Hodgkin, Relapsed or Refractory Diffuse Large B-Cell Lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Non-Hodgkin; Recurrence; Lymphoma, Large B-Cell, Diffuse | interventions — Cyclophosphamide; Doxorubicin; Vincristine; Prednisone; Rituximab

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Diffuse Large B-Cell Lymphoma (DLBCL): Participants, who were not treated previously for DLBCL, will receive rituximab (MabThera) in combination with Cyclophosphamide, Hydroxydaunorubicin, Oncovin, Prednisone (CHOP) or CHOP-like chemotherapy at the treating physician's discretion and according to package labeling, within approved indication and local approval status of respective drugs. Participants will be followed up for safety and efficacy in accordance with routine practice until progression of disease, unacceptable toxicity, withdrawal of consent or death from any reason.
  Interventions: Drug: Cyclophosphamide; Drug: Hydroxydaunorubicin; Drug: Oncovin; Drug: Prednisone; Drug: Rituximab

INTERVENTIONS:
Drug: Cyclophosphamide — Administered at the treating physician's discretion and according to package labeling, within approved indication and local approval status of the drug.
Drug: Hydroxydaunorubicin — Administered at the treating physician's discretion and according to package labeling, within approved indication and local approval status of the drug.
Drug: Oncovin — Administered at the treating physician's discretion and according to package labeling, within approved indication and local approval status of the drug.
Drug: Prednisone — Administered at the treating physician's discretion and according to package labeling, within approved indication and local approval status of the drug.
Drug: Rituximab — Administered at the treating physician's discretion and according to package labeling, within approved indication and local approval status of the drug.
  Other Names: MabThera

SUMMARY:
Evaluation of efficacy, safety profile and tolerability of rituximab (MabThera) in combination with chemotherapy in the treatment of Diffuse Large B-Cell Lymphoma (DLBCL). Participants, who were not treated previously for DLBCL, will receive MabThera in combination with Cyclophosphamide, Hydroxydaunorubicin, Oncovin, Prednisone (CHOP) or CHOP-like chemotherapy according to registered indication. Patients will be followed up for safety and efficacy evaluation in accordance with routine practice. The study will be non-interventional and by its design purely observational. All treatments prescribed during the observation period will be at the treating physician's discretion and will be prescribed according to package labeling, within approved indication and local approval status of respective drugs.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed cluster of differentiation antigen 20 (CD20) positive Diffuse Large B-Cell Lymphoma according to the World Health Organization/Revised European-American Classification of Lymphoid Neoplasms (WHO/REAL) classification
* Age > or =18 years
* Performance status < or = 2 on the Eastern Cooperative Oncology Group (ECOG) scale
* Women of child-bearing potential must agree to use effective contraception for the entire treatment period and during the 12 months thereafter

Exclusion Criteria:

* Transformed lymphoma (secondary to "low-grade" follicular lymphoma)
* Grade 1, 2 or 3a follicular lymphoma
* Primary or secondary central nervous system (CNS) involvement
* Patients with prior or concomitant malignancies except non-melanoma skin cancer or adequately treated in situ cervical cancer
* Major surgery (excluding lymph node biopsy) within 28 days prior to registration.
* Poor renal function: Serum creatinine > 2.0 mg/dl (177 micromol/L)
* Pregnancy
* Poor hepatic function: total bilirubin > 2.0 mg/dl (34 micromol/L), aspartate transaminase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) or alanine transaminase (ALT) (serum glutamic pyruvic transaminase [SGPT]) or alkaline phosphatase (AP) > 3 x the upper limit of normal unless these abnormalities are related to lymphoma.
* Known human immunodeficiency virus (HIV) infection or active viral hepatitis, specifically hepatitis B virus (HBV) or hepatitis C virus (HCV) infection.
* Serious underlying medical conditions, which could impair the ability of the patient to participate in the trial
* Life expectancy < 6 months
* Known sensitivity or allergy to murine products
* Treatment within a clinical trial within 30 days prior to trial entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with aggressive B-cell lymphoma (Diffuse Large B-Cell Lymphoma [DLBCL])
Sampling Method: Non-Probability Sample
Enrollment: 154 (Actual)
Dates: Start 2005-08; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (4):
- Serbia (4):
  - Belgrade
  - Kamenitz
  - Kragujevac
  - Niš

RESULTS

PARTICIPANT FLOW:
Groups:
- Diffuse Large B-Cell Lymphoma: Participants, who were not treated previously for diffuse large B cell lymphoma (DLBCL), and received rituximab (MabThera) in combination with Cyclophosphamide, Hydroxydaunorubicin, Oncovin, Prednisone (CHOP) or CHOP-like chemotherapy at the treating physician's discretion and according to package labeling, within approved indication and local approval status of respective drugs. Participants were followed up for safety and efficacy in accordance with routine practice until progression of disease, unacceptable toxicity, withdrawal of consent or death from any reason.
Period: Overall Study
Arm/Group | Diffuse Large B-Cell Lymphoma
Started | 154
Started Induction Therapy | 151
Completed | 104
Not Completed | 50
Not completed — Not Started Induction Therapy | 3
Not completed — Adverse Event | 1
Not completed — Death | 15
Not completed — Lack of Efficacy | 3
Not completed — Lost to Follow-up | 26
Not completed — Other | 2

BASELINE CHARACTERISTICS:
Population: Full analysis population included all participants enrolled in the study and who started induction therapy.
Groups:
- Diffuse Large B-Cell Lymphoma: Participants, who were not treated previously for DLBCL, and received rituximab in combination with CHOP or CHOP-like chemotherapy at the treating physician's discretion and according to package labeling, within approved indication and local approval status of respective drugs. Participants were followed up for safety and efficacy in accordance with routine practice until progression of disease, unacceptable toxicity, withdrawal of consent or death from any reason.
Arm/Group | Diffuse Large B-Cell Lymphoma
Number analyzed (Participants) | 151
Age, Continuous [Median (Full Range); unit: years] | 58 [19 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 61
  Male | 90

OUTCOME MEASURES:

1. Primary Outcome: Probability of Event Free Survival (EFS)
Description: EFS was calculated as the time from randomization to the date of first reported event. Events were defined as disease progression or relapse, institution of a new anticancer treatment, or death from any cause without progression.
Time Frame: Up to 41 months
Population: Full analysis population.
Measure: Number (95% Confidence Interval); unit: probability of EFS
Arm/Group | Diffuse Large B-Cell Lymphoma
Number analyzed (Participants) | 151
probability of EFS | 0.695 [0.607 to 0.796]

2. Secondary Outcome: Percentage of Participants Who Were Alive
Description: Percentage of participants with survival was calculated 41 months after the first dose of study treatment.
Time Frame: Up to 41 months
Population: Full analysis population.
Measure: Number; unit: percentage of participants
Arm/Group | Diffuse Large B-Cell Lymphoma
Number analyzed (Participants) | 151
percentage of participants | 74.4

ADVERSE EVENTS:
Time Frame: 41 Months
Description: Full analysis population.
Arm/Group | Diffuse Large B-Cell Lymphoma
Serious Adverse Events (participants affected / at risk) | 25/151
Other Adverse Events (participants affected / at risk) | 14/151
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Diffuse Large B-Cell Lymphoma (N=151)
Herpes zoster (Infections and infestations) | 1
Peritonitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Anaemia (Blood and lymphatic system disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 2
Haematotoxicity (Blood and lymphatic system disorders) | 1
Leukopenia (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 1
Haemorrhage intracranial (Nervous system disorders) | 1
Arrhythmia (Cardiac disorders) | 1
Cardiac disorder (Cardiac disorders) | 1
Cardiomyopathy (Cardiac disorders) | 1
Death (General disorders) | 1
Disease progression (General disorders) | 11
Disease recurrence (General disorders) | 3
Drug resistance (General disorders) | 1
Sudden death (General disorders) | 1
Ejection fraction decreased (Investigations) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Diffuse Large B-Cell Lymphoma (N=151)
Neutropenia (Blood and lymphatic system disorders) | 2
Headache (Nervous system disorders) | 1
Eye swelling (Eye disorders) | 1
Arrhythmia (Cardiac disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 5
Proctalgia (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 2
Chills (General disorders) | 1
Fatigue (General disorders) | 1
Pyrexia (General disorders) | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.